CLINICAL TRIAL: NCT00744029
Title: Population-Based Intervention to Reduce Prehospital Delays in Patients With Stroke and Transient Ischaemic Attack
Brief Title: Reduction of Prehospital Delays in Stroke and Transient Ischaemic Attack (TIA)
Acronym: BASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Prof. Stefan N. Willich, Institute for Social Medicine, Epidemiology and Health Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Project Z1b
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2008-09-01 (Estimated); Status verified 2008-08

CONDITIONS: Stroke
Keywords: prehospital delays; intervention; population-based; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Educational letter indicating stroke symptoms and emphasizing the importance of calling the emergency medical services (EMS) as well as a bookmark and sticker with the EMS telephone number.
  Interventions: Behavioral: educational material
- Control group (No Intervention): No intervention was performed

INTERVENTIONS:
Behavioral: educational material — Educational letter indicating stroke symptoms and emphasizing the importance of calling the emergency medical services (EMS) as well as a bookmark and sticker with the EMS telephone number.
  Arms: Intervention group

SUMMARY:
In patients with acute stroke, systemic thrombolysis needs to be administered within three hours of symptom onset. The aim of the present study was to reduce prehospital delays in a population-based intervention.The intervention consisted of an educational letter indicating stroke symptoms and emphasizing the importance of calling the emergency medical services (EMS). The investigators additionally included a bookmark and sticker with the EMS telephone number. A total of 75,720 inhabitants received the intervention. Between 2004 and 2005, 741 patients with cerebrovascular events were admitted from the control areas (n=24) and 647 from the intervention areas (n=24).

DETAILED DESCRIPTION:
Background and Purpose:

In patients with acute stroke, systemic thrombolysis needs to be administered within three hours of symptom onset. The aim of the present study was to reduce prehospital delays in a population-based intervention.

Methods:

We performed a cluster-randomized trial with 48 zip code areas as cluster units in the catchment area of three inner-city hospitals in Berlin. The primary endpoint was time between symptom onset and hospital admission. The intervention consisted of an educational letter indicating stroke symptoms and emphasizing the importance of calling the emergency medical services (EMS). We additionally included a bookmark and sticker with the EMS telephone number. We fitted a lognormal survival regression model (time-to-admission) with frailty terms shared by inhabitants of the same zip code area.

ELIGIBILITY:
Inclusion Criteria:

* All patients with stroke or transient ischaemic attacks from the postal code areas of the study being admitted to one of the participating hospitals

Exclusion Criteria:

* Patients with stroke or transient ischaemic attacks from outside the postal code areas of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1388 (Actual)
Dates: Start 2004-02; Primary Completion 2005-12 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Time between symptom onset and hospital admission | Admission to hospital

SECONDARY OUTCOMES:
Proportion of patients with thrombolysis | hospital stay
Mortality | hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Stefan N Willich, MD, Principal Investigator — Institute for Social Medicine, Epidemiology and Health Economics
Locations (1):
- Institute of Social Medicine, Epidemiology and Health Economics, Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Muller-Nordhorn J, Nolte CH, Rossnagel K, Jungehulsing GJ, Reich A, Roll S, Villringer A, Willich SN. Knowledge about risk factors for stroke: a population-based survey with 28,090 participants. Stroke. 2006 Apr;37(4):946-50. doi: 10.1161/01.STR.0000209332.96513.82. Epub 2006 Mar 2. PMID 16514090
- [Result] Rossnagel K, Jungehulsing GJ, Nolte CH, Muller-Nordhorn J, Roll S, Wegscheider K, Villringer A, Willich SN. Out-of-hospital delays in patients with acute stroke. Ann Emerg Med. 2004 Nov;44(5):476-83. doi: 10.1016/j.annemergmed.2004.06.019. PMID 15520707
- [Result] Jungehulsing GJ, Rossnagel K, Nolte CH, Muller-Nordhorn J, Roll S, Klein M, Wegscheider K, Einhaupl KM, Willich SN, Villringer A. Emergency department delays in acute stroke - analysis of time between ED arrival and imaging. Eur J Neurol. 2006 Mar;13(3):225-32. doi: 10.1111/j.1468-1331.2006.01170.x. PMID 16618337
- [Result] Jungehulsing GJ, Muller-Nordhorn J, Nolte CH, Roll S, Rossnagel K, Reich A, Wagner A, Einhaupl KM, Willich SN, Villringer A. Prevalence of stroke and stroke symptoms: a population-based survey of 28,090 participants. Neuroepidemiology. 2008;30(1):51-7. doi: 10.1159/000115750. Epub 2008 Feb 7. PMID 18259083
- [Derived] Muller-Nordhorn J, Wegscheider K, Nolte CH, Jungehulsing GJ, Rossnagel K, Reich A, Roll S, Villringer A, Willich SN. Population-based intervention to reduce prehospital delays in patients with cerebrovascular events. Arch Intern Med. 2009 Sep 14;169(16):1484-90. doi: 10.1001/archinternmed.2009.232. PMID 19752406